CLINICAL TRIAL: NCT02578875
Title: Evaluation of MiSeq for Microbial Identification in Specimens
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 160001; 16-CC-0001
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Blood Stream Infections
Keywords: Sequence Technique; Infectious Disease; Pathogen Detection; Diagnostic; Natural History
MeSH Terms: conditions — Communicable Diseases; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sample: Discarded patient samples and autopsy material

SUMMARY:
Background:

Researchers are testing a new way to find out what causes infections in people in hospitals.

Current techniques use chemical or biological tests on a person s samples. Samples are blood, tissue, stool, saliva, urine, etc. Researchers are testing new techniques that use a device called MiSeq. It can sequence all of the DNA (genetic material) in a sample. This may show microorganisms, such as bacteria, fungi, and viruses that cause infection. Researchers want to know if the new test works as well or better than current tests. They will do this by looking at about 250 samples.

Objective:

To test if MiSeq works as well as or better than current tests to identify microorganisms that cause infection.

Eligibility:

NIH patients whose samples have been sent to the Microbiology Service s lab for routine microbiologic testing.

Design:

Participants will consent to have samples they gave as part of their routine medical care used in the study. For those under age 18, a parent or legal guardian will consent.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and optimize testing that uses a next-generation DNA sequencing instrument, Illumina MiSeq, along with the associated computer infrastructure and bioinformatics software required for sequence analysis. This system is ultimately intended for use by the NIH Clinical Center Department of Laboratory Medicine to identify infectious agents in primary patient specimens. Next generation sequencing techniques based on sequencing of total DNA from primary specimens are expected to have many advantages over classical microbiological approaches. These include the detection of pathogens directly from primary specimens that may be difficult or impossible to culture.

In this study, discarded patient samples and autopsy material will be tested with the MiSeq system to identify and classify bacteria, viruses, and other pathogens. For the purpose of this study, the term samples will refer to any sample such as swabs, tissue biopsies, blood, feces, saliva, urine, wound, etc. The investigators analyzing the sequencing results will be blinded to the microbiology culture results for a validation subset of specimens to be tested with the MiSeq system. The results of the MiSeq analysis will be converted into a form that can be compared with the Microbiology Services official culture results that are stored in the laboratory information system (software from SCC SOFT Computer [Clearwater, FL, USA]).

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Discarded specimens will be used for this study.
  2. Patients from whom the specimens are derived are required to be consented.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical Center patients@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluate and optimize testing that uses a next-generation DNA sequencing instrument, Illumina MiSeq, along with the associated computer infrastructure and bioinformatics software required to sequence analysis | At study completion
  Evaluate and optimize testing that uses a next generation DNA sequencing instrument, Illumina MiSeq, along with the associated computer infrastructure and bioinformatics software required to sequence analysis

CONTACTS AND LOCATIONS:
Overall Officials: Adrian M Zelazny, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-CC-0001.html